CLINICAL TRIAL: NCT05091320
Title: Mechanical Thrombectomy of Medium Sized Vessels "M2 of MCA" :a Clinical Trial
Brief Title: Mechanical Thrombectomy of Medium Sized Vessels "M2 of MCA".
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Nageeb, assistant lecurer of neurology, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Neurointervintion and stroke
Record Dates: First submitted 2021-09-23; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Stroke, Acute Ischemic
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: case control
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mechanical thrombectomy (Active Comparator): this arm will include all patient underwent mechanical thrombectomy, either alone or after failure of medical treatment.
  Interventions: Drug: Mechanical thrombectomy; Drug: medical treatment
- medical managemnet (Active Comparator): this arm will include all patients who received medical treatment only, either anti-platelet or alteplase.
  Interventions: Drug: medical treatment

INTERVENTIONS:
Drug: Mechanical thrombectomy — Mechanical thrombectomy is interventional method and the first line management in large vessel occlusion in acute ischemic stroke
  Arms: Mechanical thrombectomy
Drug: medical treatment — medical management of patient according guide lines, either alteplase if presented in it's time window, or anti-platelet

SUMMARY:
Mechanical thrombectomy recently has revolutionized the treatment of stroke. Trials have demonstrated the superiority of mechanical thrombectomy in large vessel occlusions, such as in the intracranialinternal carotid artery and proximal, middle cerebral artery (M1), middle cerebral artery trunk (M1), have relatively high rates of revascularization and favorable clinical outcomes after MT. , However second-order branches of the middle cerebral artery (M2) occlusions (postbifurcation in the Sylvian fissure) were underrepresented or not represented in the trials. Posing a more significant technical challenge to the available endovascular devices because of the smaller size and tortuosity of these arteries and the greater likelihood of recanalization with intravenous thrombolysis, the overall risk-benefit remains uncertain.

DETAILED DESCRIPTION:
this study aims to:

1. compare efficacy of mechanical thrombectomy over medical treatment in occlusion of M2 division of MCA.
2. improve outcome of acute ischemic stroke.

The study will include all patients with AIS attending to emergency deparment with proven occlusion of M2 division of MCA, and deviding then into 2 groups:

Group 1 will receive medical treatment (rTPA if presented in the first 4 hours, and antiplatelet if passed time window for IVT) Group 2 will underwent mechanical thrombectomy (if accessible), and even after receiving medical treatment and not improved and comparing the outcomes of these 2 groups

c. Sample Size Calculation: Sample size was calculated using G*power, version 3.1.9.7. Estimation based on results of previous study which reported that, median (IQR) discharge NIHSS in mechanical thrombectomy group was 2 (0-4) compared to 1 (0-2) in medical management group giving medium effect size . With a power of 80% (using one-sided t-test, effect size = 0.65 and α of 0.5) the sample needed for the study was estimated to be 60 patients (30 in each group).

Study design:

All patients are subjected to the following: -

* Enrolled patients were admitted to stroke units or intensive care units.
* Intravenous t-PA was allowed if begun within < 4.5 hours after symptom onset.
* Thrombectomy will be performed with any FDA approved thrombectomy device by the use of local anesthesia (general anesthesia will be discouraged).

Imaging

* Patients presented with clinical picture and radiography suggestive of large vessel occlusion and who meet the proposed clinical criteria for EVT will be subjected to a comprehensive evaluation with:
* Arterial imaging of the cerebral circulation with preferably with CTA or alternatively with magnetic resonance angiography to
* Perfusion imaging with perfusion CT or with diffusion weighted imaging MRI can allow identification and quantification of the ischemic penumbra and, therefore, is useful for assessing patient eligibility for EVT in the extended time window.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Cerebral infarction in anterior circulation involving occlusion of M2 MCA, proven by CTA
* With or without IV thrombolysis
* Access to endovascular treatment within 24 hours from onset.

Exclusion Criteria:

1. Proven proximal occlusion of MCA.
2. Disability prior to the stroke (mRS >3)
3. Opposition of the patient or their family

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Clinical neurological outcome | 3 months
  Clinical neurological outcome was evaluated at discharge (within one week from onset) and at 3 months by the neurologist in charge. by using National Institutes of Health Stroke Scale (NIHSS) Good clinical outcome at discharge was defined as a NIHSS score less than or equal to 2 or a decrease in NIHSS score greater than or equal to 10 points.

SECONDARY OUTCOMES:
Functional outcome | 3 months
  Functional outcome will be assessed using Modified Rankin Scale (mRS) which measures the degree of disability after stroke.
  Good functional outcome was defined as mRS less than 2 that will be assessed at one and three moth at discharge.